CLINICAL TRIAL: NCT06133517
Title: An Open Label, Single-arm, Phase 2 Study of Perioperative Sacituzumab Govitecan in Combination With Zimberelimab and Domvanalimab for Patients With Muscle Invasive Bladder Cancer Ineligible for Cisplatin-based Chemotherapy
Brief Title: PeRioperative Immunotherapy Combined With Sacituzumab Govitecan in Muscle Invasive blAdder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación para el Progreso de la Oncología en Cantabria (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRISMA-1; 2023-504420-26-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Urothelial Bladder Carcinoma
MeSH Terms: interventions — sacituzumab govitecan; zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients who are eligible to participate in the study will receive 3 cycles of sacituzumab govitecan, zimberelimab and domvanalimab every 3 weeks prior to cystectomy, unless there are signs of unacceptable toxicity, progressive disease, or the patient requests withdrawal from the study. Patients who do not achieve a pCR or that achieving a pCR still have positive ctDNA will also complete an adjuvant phase of the study consisting of 12 additional cycles of zimberelimab and domvanalimab after cystectomy.
  Interventions: Drug: Sacituzumab govitecan; Drug: Zimberelimab; Drug: Domvanalimab

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab govitecan is administered at 10 mg/kg as an intravenous (IV) infusion on Days 1 and 8 of a 21-day cycle.
  Other Names: Trodelvy
Drug: Zimberelimab — ZIM is administered at 360 mg every 3 weeks as an intravenous (IV) infusion on Day 1 of a 21-day cycle.
Drug: Domvanalimab — DOM is administered at 1200 mg every 3 weeks as an intravenous (IV) infusion on Day 1 of a 21-day cycle.

SUMMARY:
The main objective of this trial is to evaluate the efficacy of the combo Sacituzumab govitecan (SG) + Zimberelimab (AB 122) (ZIM) + Domvanalimab (AB 154) (DOM), measured as pathologic complete response (pCR) rates, in the perioperative setting in patients with Muscle Invasive Bladder Cancer (MIBC) who are either unfit for platinum-based chemotherapy or unwilling to receive that therapy.

DETAILED DESCRIPTION:
This is an open label, multicenter, single arm, phase II clinical trial, which aims to evaluate the effects of perioperative treatment with sacituzumab govitecan, zimberelimab and domvanalimab in patients with confirmed histological diagnosis of urothelial bladder carcinoma pT2-T4a cN0-1 cM0 non-eligible or who refuse to receive cisplatin-based neoadjuvant chemotherapy.

Patients who are eligible to participate in the study will receive 3 cycles of sacituzumab govitecan, zimberelimab and domvanalimab every 3 weeks prior to cystectomy, unless there are signs of unacceptable toxicity, progressive disease or the patient requests withdrawal from the study. Patients who do not achieve a pCR or that achieving a pCR still have positive ctDNA will also complete an adjuvant phase of the study consisting of 12 additional cycles of zimberelimab and domvanalimab.

To progressively test the safety of the proposed combination, this study has been developed in two stages with the aim of preserving patient's safety as a priority. This study includes a preliminary assessment about the safety of the combinations. Thus, there will be a safety run-in period in which 8 patients will receive the SG+ZIM combination to confirm the tolerability of this doublet in patients with MIBC.

Once the safety of this doublet has been confirmed by an external safety committee then the study will proceed to an additional safety-run in cohort with the triplet.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the study procedures and requirements and restrictions in this protocol.
3. Age ≥ 18 years.
4. Muscle invasive urothelial carcinoma stage cT2-T4cN0-1cM0. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) urothelial carcinoma pattern.
5. Fit and planned for cystectomy (according to local guidelines).
6. Refusal of neoadjuvant cisplatin-based chemotherapy or patients in whom neoadjuvant cisplatin-based therapy is not appropriate. (This will be determined by the investigator and not solely based in Galsky Criteria).
7. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens (blocks preferred) or at least 15 unstained slides, with an associated pathology report, for testing at the study sponsor site. Patients with fewer than 15 unstained slides available at baseline (but no fewer than 10) may be eligible following discussion with the PI of the study.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
9. Adequate hematologic and end-organ function tests defined by the following:

   1. White Blood Cell (WBC) ≥ 2.0x109/L,
   2. Neutrophils ≥1.5x109/L,
   3. Platelets ≥100 x109/L,
   4. Hemoglobin ≥ 10 g/dL,
   5. Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation
   6. Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal(ULN),
   7. Alanine aminotransferase (ALT) ≤2.5 x ULN,
   8. Bilirubin ≤1.5 X ULN.
10. Adequate coagulation (Prothrombin Time [PT]) or International Normalized Ratio [INR] and Activated Partial Thromboplastin Time [aPTT]) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
11. Negative pregnancy test within 3 days of Day 1 Cycle 1 for female patients of childbearing potential.
12. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.

Exclusion Criteria:

1. Concurrent enrollment in another interventional clinical trial, unless in a follow-up period or it is an observational study.
2. Having received previous anticancer therapy including:

   1. Any investigational anticancer therapy received within 28 days or 5 half-lives (whichever is longer) of first dose of study treatment.
   2. Any previous intravenous chemotherapy specific for bladder cancer.
   3. Previous systemic treatment with topoisomerase 1 inhibitors.
   4. Prior Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4) or Programmed death-1(PD-1)/ programmed death-ligand 1(PD-L)1-targeting immunotherapy.
   5. Previous treatment with high dose chemotherapy and bone marrow transplant
   6. Previous radiotherapy specific for bladder cancer
3. Underlying medical conditions that might make the administration of study drugs hazardous or that might obscure the interpretation of adverse events including:

   * 3.1 Known or suspected autoimmune disease. Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus or autoimmune vasculitis (e.g., Wegener's granulomatosis) are excluded from this study; Patients with other autoimmune disorders such as a history of Hashimoto's thyroiditis [only requiring hormone replacement], type I diabetes, psoriasis [not requiring systemic treatment], or conditions not expected to recur in the absence of an external trigger are allowed to participate.
   * 3.2 History of primary immunodeficiency.
   * 3.3 A positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA), active tuberculosis, or other active infection requiring therapy at the time of inclusion.

   HIV positive patients are allowed as far as they have the disease controlled according to their treating physicians based on lymphocyte counts and viral load.

   - 3.4 Medical conditions requiring the use of immunosuppressive medications, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) will be allowed.
4. Patient receiving treatment with inhibitors or inducers of UGT1A1 at the time of enrollment.
5. Patient receiving treatment with high dose systemic corticosteroids (>10 mg of prednisone or its equivalent) within 2 weeks of C1D1.
6. Patients who have received a vaccination within 30 days prior to inclusion (examples include, but are not limited to, intranasal influenza vaccines, typhoid [oral] vaccines, and Bacillus Calmette-Guerin [BCG]). Patients are allowed to receive the COVID-19 vaccine to reduce the risk and complications of COVID-19 infection. The study visits should continue as planned if vaccination occurs while the patient is on the study.
7. Malignancy, other than urothelial cancer, in the previous 2 years. Patients with low-risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 6, and Prostatic specific antigen (PSA) ≤ 10 ng/mL) appropriately treated or that are treatment-naive and undergoing active surveillance are eligible. Also, noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin, or ductal carcinoma in situ of the breast, that have undergone potentially curative therapy are not excluded.
8. Major surgical procedure within 4 weeks prior to enrollment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis or treatment of its urothelial cancer.
9. Severe infection within 4 weeks prior to enrollment in the study including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
10. Met any of the following criteria for cardiac disease:

    1. Myocardial infarction or unstable angina pectoris within 6 months of enrollment.
    2. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication).
    3. History of QT interval prolongation.
11. Patient currently on dialysis.
12. Gastrointestinal perforation within 6 months of enrollment.
13. Patients who have organ allografts.
14. Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
15. Known allergy or hypersensitivity to study drugs formulations.
16. Patients who have invasive catheters that under the investigator criteria might put the patient at risk of developing severe complications due to neutropenia development.
17. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy measured as pathologic complete response rates of the combo SG+ZIM+DOM in the perioperative setting in patients with MIBC who are either unfit for platinum-based chemotherapy or unwilling to receive that therapy. | 42 months
  Efficacy of the combination of sacituzumab govitecan, zimberelimab and domvanalimab measured as pathologic complete response (pCR) rates.
  pCR is defined as absence of residual viable tumor (ypT0) in the radical cystectomy specimen and in the resected lymph nodes (ypN0) (post-treatment).

SECONDARY OUTCOMES:
To evaluate the downstaging rate induced by the combo | 42 months
  Downstaging is defined as any non-muscle invasive residual disease after treatment in the cystectomy specimen (i.e ypTis, ypTa,ypT1).
To measure overall survival (OS) and disease-free survival (DFS) in the study population | 42 months
  OS is defined as the time from informed consent signature to death from any cause.
To evaluate the safety of the combo | 42 months
  Safety and tolerability of the combination of sacituzumab govitecan, zimberelimab and domvanalimab measured as the incidence, nature and severity of adverse events (AEs).
To identify predictive biomarkers associated with response to SG + ZIM + DOM. | 42 months
  Cancer associated fibroblast (CAFs) as predictors of response. Immune sub-populations as predictors of response
To gain knowledge about the role of ctDNA in the perioperative setting | 42 months
  This parameter will be measured by ctDNA clearance, defined as the proportion of patients who are ctDNA positive at baseline and ctDNA negative after concluding the neoadjuvant component of the treatment, at the time of concluding neoadjuvant treatment and at the time post cystectomy.
To explore the role of adjuvant ZIM+DOM in selected patients after definitive surgical treatment | 42 months
  DFS event is defined as any of the following: development of distant metastasis of urothelial carcinoma or presence of pelvic recurrence of urothelial carcinoma (including soft tissue and regional lymph nodes) or death from any cause.
  OS is defined as the time from informed consent signature to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Duran, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla
Locations (10):
- Spain (10):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - ICO Badalona, Badalona, Barcelona
  - Hospital Duran i Reynals (ICO L´Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid, Valladolid